CLINICAL TRIAL: NCT02458079
Title: Pentoxyphilline Versus Fecal Microbiota Therapy in Severe Alcoholic Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AH-02
Record Dates: First submitted 2015-05-23; First posted 2015-05-29 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2017-07

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxiphylline (Experimental)
  Interventions: Drug: Pentoxiphylline
- Stool Microbiota Transplantation (Active Comparator)
  Interventions: Drug: Stool microbiota transplantation

INTERVENTIONS:
Drug: Pentoxiphylline
  Arms: Pentoxiphylline
Drug: Stool microbiota transplantation
  Arms: Stool Microbiota Transplantation

SUMMARY:
Treatment for severe alcoholic hepatitis patients not eligible for steroid therapy is a dilemma. Pentoxyfilline has been shown to have no improvement in outcomes as per current studies and liver transplantation is with great risk of recidivism in this difficult to treat cohort of patients. Dysbiosis forms the central role in severe alcoholic hepatitis patients and modulation of gut microbiota by way of healthy donor fecal transplantation could prove to be a novel way to treating these patients who are ineligible for standard therapy. This study utilizes correction of dysbiosis in severe alcoholic hepatitis and surveys outcomes with the same with respect to survival and liver disease severity scores.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of severe alcoholic hepatitis who are steroid ineligible, are non responders or are intolerant
* Severe alcoholic hepatitis defined as Maddrey's Discriminant Function Score (4.6 x (PT test - control))+ S.Bilirubin in mg/dl of more than 32 OR a patient of alcoholic hepatitis (defined as AST:ALT ratio > 2:1) who presents with any grade of hepatic encephalopathy
* Conventional therapy defined as oral steroid therapy (Wysolone ® 40mg once a day for 7 days)
* Failure of therapy defined as a Lille Model Score (http://www.lillemodel.com) of >0.45 at day 8 of steroid therapy OR emergence of complications of steroid therapy or intolerance to steroid protocol or ineligible for steroid therapy.
* Ineligibility for steroid therapy includes - Renal dysfunction, evidence of active sepsis or foci of sepsis, gastro intestinal bleeding and disseminated intravascular coagulation, steroid intolerance, steroid related uncontrolled hyperglycemia which precludes therapy, uncontrolled diabetes mellitus
* A Psychologist will be arranged for recipients who are on Fecal Transplant protocol for psychological support throughout the period of one week, during which the transplant procedure will be performed

  1. Healthy persons who are willing for faeces donation have to be a close family member
  2. The donor will be required to give a written consent for faeces donation
  3. Once consent is taken, the donor will have to undergo the following screening measures:

     1. Clostridium difficile toxins A and B by EIA
     2. Routine bacterial culture for enteric pathogens in stool
     3. Ova and parasites
     4. Blood serology for viruses - human immunodeficiency virus [HIV, type 1 and 2] HAV IgM, HBsAg, anti HCV Ab

Exclusion Criteria:

* Active gastrointestinal bleeding
* Intracranial bleeding
* Multi-organ failure on mechanical ventilation
* On high inotropic support
* Paralytic ileus
* Pregnancy
* Sepsis
* Failure to provide consent
* Have abnormal bowel motions
* Have abdominal complaints
* Have symptoms indicative of irritable bowel syndrome
* Have extensive travel history or predisposing factors for potentially transmittable diseases
* Have chronic alcohol intake
* Have history of substance abuse
* Are less than 18 years or more than 60 years of age
* Have HIV and Hepatitis Risk factors
* Have enteric infections
* Have inflammatory bowel disease history
* Have chronic constipation or diarrhea
* Have prior abdominal surgery or GI neoplasms
* Have Metabolic Syndrome
* Have Systemic Autoimmunity
* Have atopic diseases
* Have food and respiratory allergies
* Have any chronic pain syndromes
* Have chronic Neurologic disorders
* Have Neurodevelopmental disorders
* Have had antibiotics for any indication taken within the last 2 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Survival at 3 months | 3 months

SECONDARY OUTCOMES:
Improvement in SOFA (Sequential Organ Failure Assessment) score at 3 months | 3 month
Improvement in CTP (Child Turcotte Pugh Score) score at 3 months | 3 month
Improvement in MELD (Model for End Stage Liver Disease) score at 3 months | 3 month
Short term mortality in both groups | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India